CLINICAL TRIAL: NCT03372109
Title: A Randomized Controlled Trial to Evaluate the Effects of Repeated Periods of Modified Fasting to Support Healthy Natural Weight Management and Prevention of Weight Gain in Overweight But Generally Healthy Adults Over the Winter Holiday Period
Brief Title: Evaluate the Effects of Repeated Periods of Modified Fasting to Support Healthy Natural Weight Management and Prevention of Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CL092
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes | interventions — Geritol; Minerals; Fish Oils; Phosphatidylinositol 3-Kinases; turmeric extract; ubiquinol; Calcium; Hesperidin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Fasting Arm (Active Comparator): Dietary Supplements administered daily for 52 days with a meal replacement shake administered two days per week for the study duration
  Interventions: Dietary Supplement: Meal replacement shake; Dietary Supplement: Multivitamin and mineral capsules; Dietary Supplement: Fish oil with sesame lignans and olive extract softgel; Dietary Supplement: Prebiotic Chewable tablet; Dietary Supplement: Clove Extract and Maqui Berry extract capsule; Dietary Supplement: .Whole Food Blend capsule; Dietary Supplement: Turmeric extract capsule; Dietary Supplement: European White Kidney Bean capsule; Dietary Supplement: Saffron extract capsule; Dietary Supplement: Ubiquinol with Fulvic acid complex softgel; Dietary Supplement: Calcium with Hesperidin and gynostemma extract tablet
- Placebo (Placebo Comparator): Multivitamin tablet administered daily for 52 days
  Interventions: Dietary Supplement: Multivitamin and mineral supplement

INTERVENTIONS:
Dietary Supplement: Meal replacement shake — Meal replacement shake taken two days per week during the modified fasting periods
  Arms: Modified Fasting Arm
Dietary Supplement: Multivitamin and mineral capsules — Multivitamin/mineral supplement
  Arms: Modified Fasting Arm
Dietary Supplement: Fish oil with sesame lignans and olive extract softgel — Wild Fish Oil Concentrate 2000mg, Olive Extract 300mg, Sesame seed lignan extract 10mg/2 softgels
  Arms: Modified Fasting Arm
Dietary Supplement: Prebiotic Chewable tablet — Prebiotic Fiber 1,400 mg/tablet
  Arms: Modified Fasting Arm
Dietary Supplement: Clove Extract and Maqui Berry extract capsule — Clove extract 250mg and maqui berry extract 200mg/capsule
  Arms: Modified Fasting Arm
Dietary Supplement: .Whole Food Blend capsule — Whole food blend 1000mg/3 capsules
  Arms: Modified Fasting Arm
Dietary Supplement: Turmeric extract capsule — Turmeric 25:1 extract 400mg/capsule
  Arms: Modified Fasting Arm
Dietary Supplement: European White Kidney Bean capsule — White kidney bean extract 100mg/capsule
  Arms: Modified Fasting Arm
Dietary Supplement: Saffron extract capsule — Saffron extract 88.25mg/capsule
  Arms: Modified Fasting Arm
Dietary Supplement: Ubiquinol with Fulvic acid complex softgel — Ubiquinol 100mg and Fulvic Acid complex 100mg/softgel
  Arms: Modified Fasting Arm
Dietary Supplement: Calcium with Hesperidin and gynostemma extract tablet — Calcium 130mg. hesperidin 500mg and gynostemma extract 450mg/ tablet
  Arms: Modified Fasting Arm
Dietary Supplement: Multivitamin and mineral supplement — Multivitamin and multimineral supplement
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of repeated periods of modified fasting in support of healthy weight management and prevention of weight gain over the winter holiday period (mid-November to early January) in comparison to regular diet and activity.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled trial in which subjects assigned to the modified fasting cohort will undergo consecutive weekly cycles of modified fasting for two consecutive days.

The primary objective is to assess the effects of repeated periods of modified fasting on body weight.

The secondary objectives include assessment of the effects of modified fasting on percent body fat, waist circumference and fasting levels of hs-CRP (hs-C-reactive protein), IL-6 (Interleukin-6), IL-8 (interleukin-8), IL-12 (interleukin-12), TNF-a (tumor necrosis factor-alpha), IGF-1 (insulin-like growth factor 1), IGFBP-1 (insulin-like growth factor-binding protein 1) , Total Cholesterol, LDL cholesterol, HDL cholesterol, Glucose, Triglyceride, Insulin, Vitamin-D, 25-Hydroxy,

Participants will undergo assessments of blood tests, vital signs, BMI, body weight, waist circumference and percent body fat.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, male or female, 21-65 years of age
* A body mass index (BMI) of 23-34.9
* Generally healthy and having no significant difficulty with digestion of food
* Has been generally weight stable for the past six months
* Willing to discontinue use of any (non-study) multivitamin or Vitamin D supplements during the study
* Willing and able to give written informed consent
* Clearly understands the procedures and study requirements
* Willing and able to comply with all study procedures, including following the recommendations to maintain their usual diet and regular activity, as per protocol
* Able to communicate, including reading, in English

Primary Exclusion Criteria:

* Having smoked any cigarette, electronic cigarette, cigar, pipe, or used a recreational drug in the past 30 days
* History of allergy or sensitivity to any component of the study products including milk, soy and almonds
* Donation of blood with 30 days prior to screening/baseline
* Inability to provide a venous blood sample
* Participation in another study within 30 days prior to baseline/screening
* Being pregnant or planning on becoming pregnant during study participation; or breast feeding
* Having been diagnosed, received medical treatment or taking medication daily for the following medical condition(s):
* Diabetes mellitus
* Eating disorder
* Acute or chronic inflammatory disease or autoimmune disease
* Cardiovascular disease
* Gastrointestinal disease including gallbladder problems, gallstones or biliary tract obstruction
* Thyroid disease (unless on a stable dose of medication for 3 months prior to screening and unlikely to change medication or dose during the study)
* Hypertension (unless on a stable dose of medication for 3 months prior to screening and unlikely to change medication or dose during the study)
* Psychiatric disorder
* Neurologic condition/disease
* Cancer (unless skin cancer other than melanoma which has been treated > 3 years prior to Baseline/screening)
* Active or chronic liver, pancreatic and kidney disease
* Blood coagulation disorder
* Other condition or medication use that would preclude participation in the study in the judgment of the investigator/sub-investigator (Sub-I)
* Currently taking or having taken within the 30 days prior to screening/baseline any hormone replacement therapy (including DHEA (dehydroepiandrosterone), estrogen, progesterone, or testosterone; except those utilized as a method of birth control and which have been taken for > 3 months, with no anticipated change for the duration of the study)
* Currently taking any of the nutritional supplements used in the study and unwilling to discontinue use at least 14 days prior to screening.
* Currently taking a medication or nutritional supplement specifically for weight loss and unwilling to discontinue use 14 days prior to the first dosing of study supplements
* Currently participating in a weight loss program and unwilling to discontinue participation prior to enrollment into the study
* Currently taking an anti-coagulant, anti-platelet medication or a glucose lowering medication
* Having had a surgical procedure or having an internal medical device which, in the judgment of the PI/Sub-I, would preclude participation in the study
* Having abnormal screening laboratory test values including bilirubin > 2.5 x ULN (upper limit of normal), AST/SGOT(aspartate aminotransferase/serum glutamin oxaloacetic transaminase) and ALT/SGPT (alanine aminotransferase/serum glutamic pyruvic transaminase) > 2.5 x ULN, serum creatinine > 1.5 mg/dL, blood glucose < 85 mg/dL or > 125 mg/dL, and TSH(thyroid stimulating hormone) > 4.12 µIU/mL, or other lab test result(s) that would preclude study participation in the judgement of the PI/Sub-I
* Having blood pressure readings at Baseline/screening > 140 systolic or > 90 diastolic on two consecutive readings unless permitted to proceed to the next visit in the judgment of the PI/Sub-I
* Currently consumes more than 7 standard alcoholic drinks per week for women and 14 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
* Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges and tangelos
* Having any other circumstance that precludes study participation in the judgment of the PI/Sub-I including use of other nutritional supplements which will be evaluated on a case-by-case basis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Body weight | 52 days

SECONDARY OUTCOMES:
hs-CRP | 52 days
  hs-C-reactive protein
IL-6 | 52 days
  Interleukin-6
IL-8 | 52 days
  Interleukin-8
IL-12 | 52 days
  Interleukin-12
TNF-a | 52 days
  Tumor necrosis factor alpha
IGF-1 | 52 days
  Insulin-like growth factor 1
IGFBP-1 | 52 days
  Insulin-like growth factor binding protein 1
Total Cholesterol | 52 days
LDL-c | 52 days
  LDL Cholesterol
HDL-c | 52 days
  HDL Cholesterol
Glucose | 52 days
Triglycerides | 52 days
Insulin | 52 days
Vitamin D, 25-Hydroxy | 52 days
Percent body fat | 52 days
Waist circumference | 52 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joyal, M.D., Principal Investigator — LIfe Extension
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarado J, Schoenlau F, Leschot A, Salgad AM, Vigil Portales P. Delphinol(R) standardized maqui berry extract significantly lowers blood glucose and improves blood lipid profile in prediabetic individuals in three-month clinical trial. Panminerva Med. 2016 Sep;58(3 Suppl 1):1-6. PMID 27820958
- [Background] Alvarado JL, Leschot A, Olivera-Nappa A, Salgado AM, Rioseco H, Lyon C, Vigil P. Delphinidin-Rich Maqui Berry Extract (Delphinol(R)) Lowers Fasting and Postprandial Glycemia and Insulinemia in Prediabetic Individuals during Oral Glucose Tolerance Tests. Biomed Res Int. 2016;2016:9070537. doi: 10.1155/2016/9070537. Epub 2016 Nov 29. PMID 28025651
- [Background] Aranganathan S, Nalini N. Efficacy of the potential chemopreventive agent, hesperetin (citrus flavanone), on 1,2-dimethylhydrazine induced colon carcinogenesis. Food Chem Toxicol. 2009 Oct;47(10):2594-600. doi: 10.1016/j.fct.2009.07.019. Epub 2009 Jul 24. PMID 19632289
- [Background] Bales CW, Kraus WE. Caloric restriction: implications for human cardiometabolic health. J Cardiopulm Rehabil Prev. 2013 Jul-Aug;33(4):201-8. doi: 10.1097/HCR.0b013e318295019e. PMID 23748374
- [Background] Barger JL, Kayo T, Pugh TD, Prolla TA, Weindruch R. Short-term consumption of a resveratrol-containing nutraceutical mixture mimics gene expression of long-term caloric restriction in mouse heart. Exp Gerontol. 2008 Sep;43(9):859-66. doi: 10.1016/j.exger.2008.06.013. Epub 2008 Jul 9. PMID 18657603
- [Background] Barrett ML, Udani JK. A proprietary alpha-amylase inhibitor from white bean (Phaseolus vulgaris): a review of clinical studies on weight loss and glycemic control. Nutr J. 2011 Mar 17;10:24. doi: 10.1186/1475-2891-10-24. PMID 21414227
- [Background] Bitler C, Matt K, Irving M, et al. Olive extract supplement decreases pain and improves daily activities in adults with osteoarthritis and decreases plasma homocysteine in those with rheumatoid arthritis. Nutrition Research. 27(8):470-77.2007
- [Background] Bonakdar RA, Guarneri E. Coenzyme Q10. Am Fam Physician. 2005 Sep 15;72(6):1065-70. PMID 16190504
- [Background] Buchowski MS, Hongu N, Acra S, Wang L, Warolin J, Roberts LJ 2nd. Effect of modest caloric restriction on oxidative stress in women, a randomized trial. PLoS One. 2012;7(10):e47079. doi: 10.1371/journal.pone.0047079. Epub 2012 Oct 5. PMID 23071718
- [Background] Carai MA, Fantini N, Loi B, Colombo G, Riva A, Morazzoni P. Potential efficacy of preparations derived from Phaseolus vulgaris in the control of appetite, energy intake, and carbohydrate metabolism. Diabetes Metab Syndr Obes. 2009 Sep 7;2:145-53. doi: 10.2147/dmsott.s4236. PMID 21437128
- [Background] Carling D, Sanders MJ, Woods A. The regulation of AMP-activated protein kinase by upstream kinases. Int J Obes (Lond). 2008 Sep;32 Suppl 4:S55-9. doi: 10.1038/ijo.2008.124. PMID 18719600
- [Background] Cerda B, Ceron JJ, Tomas-Barberan FA, Espin JC. Repeated oral administration of high doses of the pomegranate ellagitannin punicalagin to rats for 37 days is not toxic. J Agric Food Chem. 2003 May 21;51(11):3493-501. doi: 10.1021/jf020842c. PMID 12744688
- [Background] Chan DC, Watts GF, Mori TA, Barrett PH, Redgrave TG, Beilin LJ. Randomized controlled trial of the effect of n-3 fatty acid supplementation on the metabolism of apolipoprotein B-100 and chylomicron remnants in men with visceral obesity. Am J Clin Nutr. 2003 Feb;77(2):300-7. doi: 10.1093/ajcn/77.2.300. PMID 12540386
- [Background] Cheng AL, Hsu CH, Lin JK, Hsu MM, Ho YF, Shen TS, Ko JY, Lin JT, Lin BR, Ming-Shiang W, Yu HS, Jee SH, Chen GS, Chen TM, Chen CA, Lai MK, Pu YS, Pan MH, Wang YJ, Tsai CC, Hsieh CY. Phase I clinical trial of curcumin, a chemopreventive agent, in patients with high-risk or pre-malignant lesions. Anticancer Res. 2001 Jul-Aug;21(4B):2895-900. PMID 11712783
- [Background] Chen HH, Chen YK, Chang HC, et al. Immunomodulatory Effects of Xylooligosaccharides. Food Science and Technology Research. 18(2):195-9. 2012.
- [Background] Cherif S, Rahal N, Haouala M, Hizaoui B, Dargouth F, Gueddiche M, Kallel Z, Balansard G, Boukef K. [A clinical trial of a titrated Olea extract in the treatment of essential arterial hypertension]. J Pharm Belg. 1996 Mar-Apr;51(2):69-71. French. PMID 8786521
- [Background] Chiranthanut N, Teekachunhatean S, Panthong A, Khonsung P, Kanjanapothi D, Lertprasertsuk N. Toxicity evaluation of standardized extract of Gynostemma pentaphyllum Makino. J Ethnopharmacol. 2013 Aug 26;149(1):228-34. doi: 10.1016/j.jep.2013.06.027. Epub 2013 Jun 21. PMID 23796877
- [Background] Coles, L.S., and Harris, S.B. Co Q-10 and lifespan extension, in: Advances in Anti-Aging Medicine, Vol 1, by R. Klatz, Mary Ann Liebert, Inc., Larchmont, New York, 1996
- [Background] Conley M, Le Fevre L, Haywood C, Proietto J. Is two days of intermittent energy restriction per week a feasible weight loss approach in obese males? A randomised pilot study. Nutr Diet. 2018 Feb;75(1):65-72. doi: 10.1111/1747-0080.12372. Epub 2017 Aug 9. PMID 28791787
- [Background] D'Argenio G, Mazzacca G. Short-chain fatty acid in the human colon. Relation to inflammatory bowel diseases and colon cancer. Adv Exp Med Biol. 1999;472:149-58. doi: 10.1007/978-1-4757-3230-6_13. PMID 10736623
- [Background] Davinelli S, Bertoglio JC, Zarrelli A, Pina R, Scapagnini G. A Randomized Clinical Trial Evaluating the Efficacy of an Anthocyanin-Maqui Berry Extract (Delphinol(R)) on Oxidative Stress Biomarkers. J Am Coll Nutr. 2015;34 Suppl 1:28-33. doi: 10.1080/07315724.2015.1080108. PMID 26400431
- [Background] de Bock M, Derraik JG, Brennan CM, Biggs JB, Morgan PE, Hodgkinson SC, Hofman PL, Cutfield WS. Olive (Olea europaea L.) leaf polyphenols improve insulin sensitivity in middle-aged overweight men: a randomized, placebo-controlled, crossover trial. PLoS One. 2013;8(3):e57622. doi: 10.1371/journal.pone.0057622. Epub 2013 Mar 13. PMID 23516412
- [Background] de Vries W, Stouthamer AH. Pathway of glucose fermentation in relation to the taxonomy of bifidobacteria. J Bacteriol. 1967 Feb;93(2):574-6. doi: 10.1128/jb.93.2.574-576.1967. PMID 6020562
- [Background] Duenas M, Munoz-Gonzalez I, Cueva C, Jimenez-Giron A, Sanchez-Patan F, Santos-Buelga C, Moreno-Arribas MV, Bartolome B. A survey of modulation of gut microbiota by dietary polyphenols. Biomed Res Int. 2015;2015:850902. doi: 10.1155/2015/850902. Epub 2015 Feb 22. PMID 25793210
- [Background] El-Marasy SA, Abdallah HM, El-Shenawy SM, El-Khatib AS, El-Shabrawy OA, Kenawy SA. Anti-depressant effect of hesperidin in diabetic rats. Can J Physiol Pharmacol. 2014 Nov;92(11):945-52. doi: 10.1139/cjpp-2014-0281. Epub 2014 Sep 19. PMID 25358020
- [Background] Ershler WB, Sun WH, Binkley N, Gravenstein S, Volk MJ, Kamoske G, Klopp RG, Roecker EB, Daynes RA, Weindruch R. Interleukin-6 and aging: blood levels and mononuclear cell production increase with advancing age and in vitro production is modifiable by dietary restriction. Lymphokine Cytokine Res. 1993 Aug;12(4):225-30. PMID 8218595
- [Background] Esposito K, Kastorini CM, Panagiotakos DB, Giugliano D. Mediterranean diet and weight loss: meta-analysis of randomized controlled trials. Metab Syndr Relat Disord. 2011 Feb;9(1):1-12. doi: 10.1089/met.2010.0031. Epub 2010 Oct 25. PMID 20973675
- [Background] Fantini N, Cabras C, Lobina C, Colombo G, Gessa GL, Riva A, Donzelli F, Morazzoni P, Bombardelli E, Carai MA. Reducing effect of a Phaseolus vulgaris dry extract on food intake, body weight, and glycemia in rats. J Agric Food Chem. 2009 Oct 14;57(19):9316-23. doi: 10.1021/jf900711z. PMID 19731962
- [Background] Garg A, Garg S, Zaneveld LJ, Singla AK. Chemistry and pharmacology of the Citrus bioflavonoid hesperidin. Phytother Res. 2001 Dec;15(8):655-69. doi: 10.1002/ptr.1074. PMID 11746857
- [Background] Gauhar R, Hwang SL, Jeong SS, Kim JE, Song H, Park DC, Song KS, Kim TY, Oh WK, Huh TL. Heat-processed Gynostemma pentaphyllum extract improves obesity in ob/ob mice by activating AMP-activated protein kinase. Biotechnol Lett. 2012 Sep;34(9):1607-16. doi: 10.1007/s10529-012-0944-1. Epub 2012 May 11. PMID 22576281
- [Background] Ghasemi T, Abnous K, Vahdati F, Mehri S, Razavi BM, Hosseinzadeh H. Antidepressant Effect of Crocus sativus Aqueous Extract and its Effect on CREB, BDNF, and VGF Transcript and Protein Levels in Rat Hippocampus. Drug Res (Stuttg). 2015 Jul;65(7):337-43. doi: 10.1055/s-0034-1371876. Epub 2014 Apr 2. PMID 24696423
- [Background] Gout B, Bourges C, Paineau-Dubreuil S. Satiereal, a Crocus sativus L extract, reduces snacking and increases satiety in a randomized placebo-controlled study of mildly overweight, healthy women. Nutr Res. 2010 May;30(5):305-13. doi: 10.1016/j.nutres.2010.04.008. PMID 20579522
- [Background] Griffin MD, Sanders TA, Davies IG, Morgan LM, Millward DJ, Lewis F, Slaughter S, Cooper JA, Miller GJ, Griffin BA. Effects of altering the ratio of dietary n-6 to n-3 fatty acids on insulin sensitivity, lipoprotein size, and postprandial lipemia in men and postmenopausal women aged 45-70 y: the OPTILIP Study. Am J Clin Nutr. 2006 Dec;84(6):1290-8. doi: 10.1093/ajcn/84.6.1290. PMID 17158408
- [Background] Handler N, Jaeger W, Puschacher H, Leisser K, Erker T. Synthesis of novel curcumin analogues and their evaluation as selective cyclooxygenase-1 (COX-1) inhibitors. Chem Pharm Bull (Tokyo). 2007 Jan;55(1):64-71. doi: 10.1248/cpb.55.64. PMID 17202703
- [Background] Hansen CH, Frokiaer H, Christensen AG, Bergstrom A, Licht TR, Hansen AK, Metzdorff SB. Dietary xylooligosaccharide downregulates IFN-gamma and the low-grade inflammatory cytokine IL-1beta systemically in mice. J Nutr. 2013 Apr;143(4):533-40. doi: 10.3945/jn.112.172361. Epub 2013 Feb 20. PMID 23427328
- [Background] Hardie DG. AMP-activated protein kinase: a key system mediating metabolic responses to exercise. Med Sci Sports Exerc. 2004 Jan;36(1):28-34. doi: 10.1249/01.MSS.0000106171.38299.64. PMID 14707764
- [Background] Hardie DG. AMPK: a key regulator of energy balance in the single cell and the whole organism. Int J Obes (Lond). 2008 Sep;32 Suppl 4:S7-12. doi: 10.1038/ijo.2008.116. PMID 18719601
- [Background] Hardie DG, Ross FA, Hawley SA. AMPK: a nutrient and energy sensor that maintains energy homeostasis. Nat Rev Mol Cell Biol. 2012 Mar 22;13(4):251-62. doi: 10.1038/nrm3311. PMID 22436748
- [Background] Hardie DG. Sensing of energy and nutrients by AMP-activated protein kinase. Am J Clin Nutr. 2011 Apr;93(4):891S-6. doi: 10.3945/ajcn.110.001925. Epub 2011 Feb 16. PMID 21325438
- [Background] Hausenblas HA, Heekin K, Mutchie HL, Anton S. A systematic review of randomized controlled trials examining the effectiveness of saffron (Crocus sativus L.) on psychological and behavioral outcomes. J Integr Med. 2015 Jul;13(4):231-40. doi: 10.1016/S2095-4964(15)60176-5. PMID 26165367
- [Background] Hausenblas HA, Saha D, Dubyak PJ, Anton SD. Saffron (Crocus sativus L.) and major depressive disorder: a meta-analysis of randomized clinical trials. J Integr Med. 2013 Nov;11(6):377-83. doi: 10.3736/jintegrmed2013056. PMID 24299602
- [Background] Heilbronn LK, Clifton PM. C-reactive protein and coronary artery disease: influence of obesity, caloric restriction and weight loss. J Nutr Biochem. 2002 Jun;13(6):316-321. doi: 10.1016/s0955-2863(02)00187-0. PMID 12088796
- [Background] Henke BR, Sparks SM. Glycogen phosphorylase inhibitors. Mini Rev Med Chem. 2006 Aug;6(8):845-57. doi: 10.2174/138955706777934991. PMID 16918491
- [Background] Hidalgo J, Flores C, Hidalgo MA, Perez M, Yanez A, Quinones L, Caceres DD, Burgos RA. Delphinol(R) standardized maqui berry extract reduces postprandial blood glucose increase in individuals with impaired glucose regulation by novel mechanism of sodium glucose cotransporter inhibition. Panminerva Med. 2014 Jun;56(2 Suppl 3):1-7. PMID 24861886
- [Background] Hokayem M, Blond E, Vidal H, Lambert K, Meugnier E, Feillet-Coudray C, Coudray C, Pesenti S, Luyton C, Lambert-Porcheron S, Sauvinet V, Fedou C, Brun JF, Rieusset J, Bisbal C, Sultan A, Mercier J, Goudable J, Dupuy AM, Cristol JP, Laville M, Avignon A. Grape polyphenols prevent fructose-induced oxidative stress and insulin resistance in first-degree relatives of type 2 diabetic patients. Diabetes Care. 2013 Jun;36(6):1454-61. doi: 10.2337/dc12-1652. Epub 2012 Dec 28. PMID 23275372
- [Background] Hosoe K, Kitano M, Kishida H, Kubo H, Fujii K, Kitahara M. Study on safety and bioavailability of ubiquinol (Kaneka QH) after single and 4-week multiple oral administration to healthy volunteers. Regul Toxicol Pharmacol. 2007 Feb;47(1):19-28. doi: 10.1016/j.yrtph.2006.07.001. Epub 2006 Aug 21. PMID 16919858
- [Background] Hosseini B, Saedisomeolia A, Wood LG, Yaseri M, Tavasoli S. Effects of pomegranate extract supplementation on inflammation in overweight and obese individuals: A randomized controlled clinical trial. Complement Ther Clin Pract. 2016 Feb;22:44-50. doi: 10.1016/j.ctcp.2015.12.003. Epub 2015 Dec 12. PMID 26850805
- [Background] Huyen VT, Phan DV, Thang P, Hoa NK, Ostenson CG. Antidiabetic effect of Gynostemma pentaphyllum tea in randomly assigned type 2 diabetic patients. Horm Metab Res. 2010 May;42(5):353-7. doi: 10.1055/s-0030-1248298. Epub 2010 Mar 8. PMID 20213586
- [Background] Ikematsu H, Nakamura K, Harashima S, Fujii K, Fukutomi N. Safety assessment of coenzyme Q10 (Kaneka Q10) in healthy subjects: a double-blind, randomized, placebo-controlled trial. Regul Toxicol Pharmacol. 2006 Apr;44(3):212-8. doi: 10.1016/j.yrtph.2005.12.002. Epub 2006 Jan 23. PMID 16431002
- [Background] Jain I, Kumar V, Satyanarayana T. Xylooligosaccharides: an economical prebiotic from agroresidues and their health benefits. Indian J Exp Biol. 2015 Mar;53(3):131-42. PMID 25872243
- [Background] NM J, RM R, G G, Maliakel B, D S, IM K. Beyond the flavour: a de-flavoured polyphenol rich extract of clove buds (Syzygium aromaticum L) as a novel dietary antioxidant ingredient. Food Funct. 2015 Oct;6(10):3373-82. doi: 10.1039/c5fo00682a. PMID 26273738
- [Background] Kaats GR, Miller H, Preuss HG, Stohs SJ. A 60day double-blind, placebo-controlled safety study involving Citrus aurantium (bitter orange) extract. Food Chem Toxicol. 2013 May;55:358-62. doi: 10.1016/j.fct.2013.01.013. Epub 2013 Jan 25. PMID 23354394
- [Background] Kato M, Tani T, Terahara N, Tsuda T. The Anthocyanin Delphinidin 3-Rutinoside Stimulates Glucagon-Like Peptide-1 Secretion in Murine GLUTag Cell Line via the Ca2+/Calmodulin-Dependent Kinase II Pathway. PLoS One. 2015 May 11;10(5):e0126157. doi: 10.1371/journal.pone.0126157. eCollection 2015. PMID 25962102
- [Background] Kamaraj S, Ramakrishnan G, Anandakumar P, Jagan S, Devaki T. Antioxidant and anticancer efficacy of hesperidin in benzo(a)pyrene induced lung carcinogenesis in mice. Invest New Drugs. 2009 Jun;27(3):214-22. doi: 10.1007/s10637-008-9159-7. Epub 2008 Aug 13. PMID 18704264
- [Background] Khanna D, Sethi G, Ahn KS, Pandey MK, Kunnumakkara AB, Sung B, Aggarwal A, Aggarwal BB. Natural products as a gold mine for arthritis treatment. Curr Opin Pharmacol. 2007 Jun;7(3):344-51. doi: 10.1016/j.coph.2007.03.002. Epub 2007 May 1. PMID 17475558
- [Background] Khoo J, Piantadosi C, Duncan R, Worthley SG, Jenkins A, Noakes M, Worthley MI, Lange K, Wittert GA. Comparing effects of a low-energy diet and a high-protein low-fat diet on sexual and endothelial function, urinary tract symptoms, and inflammation in obese diabetic men. J Sex Med. 2011 Oct;8(10):2868-75. doi: 10.1111/j.1743-6109.2011.02417.x. Epub 2011 Aug 5. PMID 21819545
- [Background] Khurana S, Venkataraman K, Hollingsworth A, Piche M, Tai TC. Polyphenols: benefits to the cardiovascular system in health and in aging. Nutrients. 2013 Sep 26;5(10):3779-827. doi: 10.3390/nu5103779. PMID 24077237
- [Background] Kim JY, Jung KJ, Choi JS, Chung HY. Modulation of the age-related nuclear factor-kappaB (NF-kappaB) pathway by hesperetin. Aging Cell. 2006 Oct;5(5):401-11. doi: 10.1111/j.1474-9726.2006.00233.x. Epub 2006 Aug 25. PMID 16939486
- [Background] Kim YJ, Kim HJ, No JK, Chung HY, Fernandes G. Anti-inflammatory action of dietary fish oil and calorie restriction. Life Sci. 2006 Apr 18;78(21):2523-32. doi: 10.1016/j.lfs.2005.10.034. Epub 2006 Jan 24. PMID 16438990
- [Background] Kleemann R, van Erk M, Verschuren L, van den Hoek AM, Koek M, Wielinga PY, Jie A, Pellis L, Bobeldijk-Pastorova I, Kelder T, Toet K, Wopereis S, Cnubben N, Evelo C, van Ommen B, Kooistra T. Time-resolved and tissue-specific systems analysis of the pathogenesis of insulin resistance. PLoS One. 2010 Jan 21;5(1):e8817. doi: 10.1371/journal.pone.0008817. PMID 20098690
- [Background] Komaroff AL. The Microbiome and Risk for Obesity and Diabetes. JAMA. 2017 Jan 24;317(4):355-356. doi: 10.1001/jama.2016.20099. No abstract available. PMID 28006047
- [Background] Lee SH, Min KJ. Caloric restriction and its mimetics. BMB Rep. 2013 Apr;46(4):181-7. doi: 10.5483/bmbrep.2013.46.4.033. PMID 23615258
- [Background] Li C, Schluesener H. Health-promoting effects of the citrus flavanone hesperidin. Crit Rev Food Sci Nutr. 2017 Feb 11;57(3):613-631. doi: 10.1080/10408398.2014.906382. PMID 25675136
- [Background] Li JJ, Huang CJ, Xie D. Anti-obesity effects of conjugated linoleic acid, docosahexaenoic acid, and eicosapentaenoic acid. Mol Nutr Food Res. 2008 Jun;52(6):631-45. doi: 10.1002/mnfr.200700399. PMID 18306430
- [Background] Li M, Lin XF, Lu J, Zhou BR, Luo D. Hesperidin ameliorates UV radiation-induced skin damage by abrogation of oxidative stress and inflammatory in HaCaT cells. J Photochem Photobiol B. 2016 Dec;165:240-245. doi: 10.1016/j.jphotobiol.2016.10.037. Epub 2016 Nov 1. PMID 27816646
- [Background] Li R, Li J, Cai L, Hu CM, Zhang L. Suppression of adjuvant arthritis by hesperidin in rats and its mechanisms. J Pharm Pharmacol. 2008 Feb;60(2):221-8. doi: 10.1211/jpp.60.2.0011. PMID 18237470
- [Background] Lin-Na S, Yong-Xiu S. Effects of polysaccharides from Gynostemma pentaphyllum (Thunb.), Makino on physical fatigue. Afr J Tradit Complement Altern Med. 2014 Apr 3;11(3):112-7. doi: 10.4314/ajtcam.v11i3.17. eCollection 2014. PMID 25371572
- [Background] Longo VD, Mattson MP. Fasting: molecular mechanisms and clinical applications. Cell Metab. 2014 Feb 4;19(2):181-92. doi: 10.1016/j.cmet.2013.12.008. Epub 2014 Jan 16. PMID 24440038
- [Background] Mace, A.E. (1964), Sample Size Determination, New York: Reinhold Publishing Corporation
- [Background] Marin YE, Wall BA, Wang S, Namkoong J, Martino JJ, Suh J, Lee HJ, Rabson AB, Yang CS, Chen S, Ryu JH. Curcumin downregulates the constitutive activity of NF-kappaB and induces apoptosis in novel mouse melanoma cells. Melanoma Res. 2007 Oct;17(5):274-83. doi: 10.1097/CMR.0b013e3282ed3d0e. PMID 17885582
- [Background] Marino G, Pietrocola F, Madeo F, Kroemer G. Caloric restriction mimetics: natural/physiological pharmacological autophagy inducers. Autophagy. 2014;10(11):1879-82. doi: 10.4161/auto.36413. PMID 25484097
- [Background] Martini C, Pallottini V, De Marinis E, Marino M, Cavallini G, Donati A, Straniero S, Trentalance A. Omega-3 as well as caloric restriction prevent the age-related modifications of cholesterol metabolism. Mech Ageing Dev. 2008 Dec;129(12):722-7. doi: 10.1016/j.mad.2008.09.010. Epub 2008 Sep 26. PMID 18930075
- [Background] Merry BJ. Molecular mechanisms linking calorie restriction and longevity. Int J Biochem Cell Biol. 2002 Nov;34(11):1340-54. doi: 10.1016/s1357-2725(02)00038-9. PMID 12200030
- [Background] Meydani M, Hasan ST. Dietary polyphenols and obesity. Nutrients. 2010 Jul;2(7):737-51. doi: 10.3390/nu2070737. Epub 2010 Jul 8. PMID 22254051
- [Background] Meyer OC. Safety and security of Daflon 500 mg in venous insufficiency and in hemorrhoidal disease. Angiology. 1994 Jun;45(6 Pt 2):579-84. doi: 10.1177/000331979404500614. PMID 8203791
- [Background] Meyer TE, Kovacs SJ, Ehsani AA, Klein S, Holloszy JO, Fontana L. Long-term caloric restriction ameliorates the decline in diastolic function in humans. J Am Coll Cardiol. 2006 Jan 17;47(2):398-402. doi: 10.1016/j.jacc.2005.08.069. PMID 16412867
- [Background] Mishra R, Joshi D. Jiao Gu Lan (Gynostemma pentaphyllum): The Chinese Rasayan-Current Research Scenario. International Journal of Research in Pharmaceutical and Biomedical Sciences. 2(4): 1483-1502, 2011.
- [Background] Miwa Y, Yamada M, Sunayama T, Mitsuzumi H, Tsuzaki Y, Chaen H, Mishima Y, Kibata M. Effects of glucosyl hesperidin on serum lipids in hyperlipidemic subjects: preferential reduction in elevated serum triglyceride level. J Nutr Sci Vitaminol (Tokyo). 2004 Jun;50(3):211-8. doi: 10.3177/jnsv.50.211. PMID 15386934
- [Background] Modaghegh MH, Shahabian M, Esmaeili HA, Rajbai O, Hosseinzadeh H. Safety evaluation of saffron (Crocus sativus) tablets in healthy volunteers. Phytomedicine. 2008 Dec;15(12):1032-7. doi: 10.1016/j.phymed.2008.06.003. Epub 2008 Aug 6. PMID 18693099
- [Background] Mostoslavsky R, Chua KF, Lombard DB, Pang WW, Fischer MR, Gellon L, Liu P, Mostoslavsky G, Franco S, Murphy MM, Mills KD, Patel P, Hsu JT, Hong AL, Ford E, Cheng HL, Kennedy C, Nunez N, Bronson R, Frendewey D, Auerbach W, Valenzuela D, Karow M, Hottiger MO, Hursting S, Barrett JC, Guarente L, Mulligan R, Demple B, Yancopoulos GD, Alt FW. Genomic instability and aging-like phenotype in the absence of mammalian SIRT6. Cell. 2006 Jan 27;124(2):315-29. doi: 10.1016/j.cell.2005.11.044. PMID 16439206
- [Background] Nielsen IL, Chee WS, Poulsen L, Offord-Cavin E, Rasmussen SE, Frederiksen H, Enslen M, Barron D, Horcajada MN, Williamson G. Bioavailability is improved by enzymatic modification of the citrus flavonoid hesperidin in humans: a randomized, double-blind, crossover trial. J Nutr. 2006 Feb;136(2):404-8. doi: 10.1093/jn/136.2.404. PMID 16424119
- [Background] Ohara T, Muroyama K, Yamamoto Y, Murosaki S. Oral intake of a combination of glucosyl hesperidin and caffeine elicits an anti-obesity effect in healthy, moderately obese subjects: a randomized double-blind placebo-controlled trial. Nutr J. 2016 Jan 19;15:6. doi: 10.1186/s12937-016-0123-7. PMID 26786000
- [Background] Palit S, Kar S, Sharma G, Das PK. Hesperetin Induces Apoptosis in Breast Carcinoma by Triggering Accumulation of ROS and Activation of ASK1/JNK Pathway. J Cell Physiol. 2015 Aug;230(8):1729-39. doi: 10.1002/jcp.24818. PMID 25204891
- [Background] Park C, Moon DO, Choi IW, Choi BT, Nam TJ, Rhu CH, Kwon TK, Lee WH, Kim GY, Choi YH. Curcumin induces apoptosis and inhibits prostaglandin E(2) production in synovial fibroblasts of patients with rheumatoid arthritis. Int J Mol Med. 2007 Sep;20(3):365-72. PMID 17671742
- [Background] Pathak N, Rai AK, Kumari R, Bhat KV. Value addition in sesame: A perspective on bioactive components for enhancing utility and profitability. Pharmacogn Rev. 2014 Jul;8(16):147-55. doi: 10.4103/0973-7847.134249. PMID 25125886
- [Background] Pazoki-Toroudi H, Amani H, Ajami M, Nabavi SF, Braidy N, Kasi PD, Nabavi SM. Targeting mTOR signaling by polyphenols: A new therapeutic target for ageing. Ageing Res Rev. 2016 Nov;31:55-66. doi: 10.1016/j.arr.2016.07.004. Epub 2016 Jul 21. PMID 27453478
- [Background] Phillips T, Leeuwenburgh C. Muscle fiber specific apoptosis and TNF-alpha signaling in sarcopenia are attenuated by life-long calorie restriction. FASEB J. 2005 Apr;19(6):668-70. doi: 10.1096/fj.04-2870fje. Epub 2005 Jan 21. PMID 15665035
- [Background] Pokusaeva K, Fitzgerald GF, van Sinderen D. Carbohydrate metabolism in Bifidobacteria. Genes Nutr. 2011 Aug;6(3):285-306. doi: 10.1007/s12263-010-0206-6. Epub 2011 Feb 16. PMID 21484167
- [Background] Poudyal H, Campbell F, Brown L. Olive leaf extract attenuates cardiac, hepatic, and metabolic changes in high carbohydrate-, high fat-fed rats. J Nutr. 2010 May;140(5):946-53. doi: 10.3945/jn.109.117812. Epub 2010 Mar 24. PMID 20335636
- [Background] Ray S, Bagchi D, Lim PM, Bagchi M, Gross SM, Kothari SC, Preuss HG, Stohs SJ. Acute and long-term safety evaluation of a novel IH636 grape seed proanthocyanidin extract. Res Commun Mol Pathol Pharmacol. 2001 Mar-Apr;109(3-4):165-97. PMID 11758648
- [Background] Razmovski-Naumovski V, Hsun-Wei Huang T, Tran V, et al. Chemistry and pharmacology of Gynostemma pentaphyllum. Phytochemistry Reviews 4:197-219, 2005
- [Background] Renny RM, Gopakumar G, Mohanan R, et al. Clove bud polyphenols (Clovinol®) reduces hangover and helps faster clearance of acetaldehyde by maintaining endogenous antioxidants and reducing inflammation: A randomized, double-blind, placebo-controlled crossover study. Under Review - Pharmacology Biochemistry & Behavior. 2016.
- [Background] Rizza S, Muniyappa R, Iantorno M, Kim JA, Chen H, Pullikotil P, Senese N, Tesauro M, Lauro D, Cardillo C, Quon MJ. Citrus polyphenol hesperidin stimulates production of nitric oxide in endothelial cells while improving endothelial function and reducing inflammatory markers in patients with metabolic syndrome. J Clin Endocrinol Metab. 2011 May;96(5):E782-92. doi: 10.1210/jc.2010-2879. Epub 2011 Feb 23. PMID 21346065
- [Background] Rojo LE, Ribnicky D, Logendra S, Poulev A, Rojas-Silva P, Kuhn P, Dorn R, Grace MH, Lila MA, Raskin I. In Vitro and in Vivo Anti-Diabetic Effects of Anthocyanins from Maqui Berry (Aristotelia chilensis). Food Chem. 2012 Mar 15;131(2):387-396. doi: 10.1016/j.foodchem.2011.08.066. PMID 26279603
- [Background] Roohbakhsh A, Parhiz H, Soltani F, Rezaee R, Iranshahi M. Molecular mechanisms behind the biological effects of hesperidin and hesperetin for the prevention of cancer and cardiovascular diseases. Life Sci. 2015 Mar 1;124:64-74. doi: 10.1016/j.lfs.2014.12.030. Epub 2015 Jan 24. PMID 25625242
- [Background] Ruth MR, Port AM, Shah M, Bourland AC, Istfan NW, Nelson KP, Gokce N, Apovian CM. Consuming a hypocaloric high fat low carbohydrate diet for 12 weeks lowers C-reactive protein, and raises serum adiponectin and high density lipoprotein-cholesterol in obese subjects. Metabolism. 2013 Dec;62(12):1779-87. doi: 10.1016/j.metabol.2013.07.006. Epub 2013 Sep 26. PMID 24075505
- [Background] Sanae F, Kamiyama O, Ikeda-Obatake K, Higashi Y, Asano N, Adachi I, Kato A. Effects of eugenol-reduced clove extract on glycogen phosphorylase b and the development of diabetes in db/db mice. Food Funct. 2014 Feb;5(2):214-9. doi: 10.1039/c3fo60514k. PMID 24336787
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Background] Shehata AS, Amer MG, Abd El-Haleem MR, Karam RA. The ability of hesperidin compared to that of insulin for preventing osteoporosis induced by type I diabetes in young male albino rats: A histological and biochemical study. Exp Toxicol Pathol. 2017 Apr 4;69(4):203-212. doi: 10.1016/j.etp.2017.01.008. Epub 2017 Jan 26. PMID 28132802
- [Background] Shults CW, Oakes D, Kieburtz K, Beal MF, Haas R, Plumb S, Juncos JL, Nutt J, Shoulson I, Carter J, Kompoliti K, Perlmutter JS, Reich S, Stern M, Watts RL, Kurlan R, Molho E, Harrison M, Lew M; Parkinson Study Group. Effects of coenzyme Q10 in early Parkinson disease: evidence of slowing of the functional decline. Arch Neurol. 2002 Oct;59(10):1541-50. doi: 10.1001/archneur.59.10.1541. PMID 12374491
- [Background] Spadafranca A, Rinelli S, Riva A, Morazzoni P, Magni P, Bertoli S, Battezzati A. Phaseolus vulgaris extract affects glycometabolic and appetite control in healthy human subjects. Br J Nutr. 2013 May 28;109(10):1789-95. doi: 10.1017/S0007114512003741. Epub 2012 Oct 9. PMID 23046862
- [Background] Taghizadeh M, Farzin N, Taheri S, Mahlouji M, Akbari H, Karamali F, Asemi Z. The Effect of Dietary Supplements Containing Green Tea, Capsaicin and Ginger Extracts on Weight Loss and Metabolic Profiles in Overweight Women: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Ann Nutr Metab. 2017;70(4):277-285. doi: 10.1159/000471889. Epub 2017 Jun 9. PMID 28595182
- [Background] Tomimori N, Tanaka Y, Kitagawa Y, Fujii W, Sakakibara Y, Shibata H. Pharmacokinetics and safety of the sesame lignans, sesamin and episesamin, in healthy subjects. Biopharm Drug Dispos. 2013 Nov;34(8):462-73. doi: 10.1002/bdd.1862. Epub 2013 Oct 17. PMID 24014208
- [Background] Umeno A, Horie M, Murotomi K, Nakajima Y, Yoshida Y. Antioxidative and Antidiabetic Effects of Natural Polyphenols and Isoflavones. Molecules. 2016 May 30;21(6):708. doi: 10.3390/molecules21060708. PMID 27248987
- [Background] Ungvari Z, Parrado-Fernandez C, Csiszar A, de Cabo R. Mechanisms underlying caloric restriction and lifespan regulation: implications for vascular aging. Circ Res. 2008 Mar 14;102(5):519-28. doi: 10.1161/CIRCRESAHA.107.168369. PMID 18340017
- [Background] Vallianou NG, Evangelopoulos A, Schizas N, Kazazis C. Potential anticancer properties and mechanisms of action of curcumin. Anticancer Res. 2015 Feb;35(2):645-51. PMID 25667441
- [Background] Varady KA, Bhutani S, Klempel MC, Kroeger CM, Trepanowski JF, Haus JM, Hoddy KK, Calvo Y. Alternate day fasting for weight loss in normal weight and overweight subjects: a randomized controlled trial. Nutr J. 2013 Nov 12;12(1):146. doi: 10.1186/1475-2891-12-146. PMID 24215592
- [Background] Verdery RB, Walford RL. Changes in plasma lipids and lipoproteins in humans during a 2-year period of dietary restriction in Biosphere 2. Arch Intern Med. 1998 Apr 27;158(8):900-6. doi: 10.1001/archinte.158.8.900. PMID 9570177
- [Background] Visnagri A, Kandhare AD, Chakravarty S, Ghosh P, Bodhankar SL. Hesperidin, a flavanoglycone attenuates experimental diabetic neuropathy via modulation of cellular and biochemical marker to improve nerve functions. Pharm Biol. 2014 Jul;52(7):814-28. doi: 10.3109/13880209.2013.870584. Epub 2014 Feb 21. PMID 24559476
- [Background] Wang M, Wang F, Wang Y, Ma X, Zhao M, Zhao C. Metabonomics study of the therapeutic mechanism of Gynostemma pentaphyllum and atorvastatin for hyperlipidemia in rats. PLoS One. 2013 Nov 1;8(11):e78731. doi: 10.1371/journal.pone.0078731. eCollection 2013. PMID 24223845
- [Background] Westphal S, Orth M, Ambrosch A, Osmundsen K, Luley C. Postprandial chylomicrons and VLDLs in severe hypertriacylglycerolemia are lowered more effectively than are chylomicron remnants after treatment with n-3 fatty acids. Am J Clin Nutr. 2000 Apr;71(4):914-20. doi: 10.1093/ajcn/71.4.914. PMID 10731497
- [Background] Witte AV, Fobker M, Gellner R, Knecht S, Floel A. Caloric restriction improves memory in elderly humans. Proc Natl Acad Sci U S A. 2009 Jan 27;106(4):1255-60. doi: 10.1073/pnas.0808587106. Epub 2009 Jan 26. PMID 19171901
- [Background] Wu X, Xiaofeng X, Shen J, Perricone NV, Preuss HG. Enhanced weight loss from a dietary supplement containing standardized Phaseolus vulgaris extract in overweight men and women. Methods (San Diego, Calif.). 12(13):15-22. 2010.
- [Background] Xiao L, Ning J, Xu G. Application of Xylo-oligosaccharide in modifying human intestinal function. African Journal of Microbiology Research. (9):2116-9, 2012.
- [Background] Yanovski JA, Yanovski SZ, Sovik KN, Nguyen TT, O'Neil PM, Sebring NG. A prospective study of holiday weight gain. N Engl J Med. 2000 Mar 23;342(12):861-7. doi: 10.1056/NEJM200003233421206. PMID 10727591
- [Background] Zamora-Ros R, Knaze V, Rothwell JA, Hemon B, Moskal A, Overvad K, Tjonneland A, Kyro C, Fagherazzi G, Boutron-Ruault MC, Touillaud M, Katzke V, Kuhn T, Boeing H, Forster J, Trichopoulou A, Valanou E, Peppa E, Palli D, Agnoli C, Ricceri F, Tumino R, de Magistris MS, Peeters PH, Bueno-de-Mesquita HB, Engeset D, Skeie G, Hjartaker A, Menendez V, Agudo A, Molina-Montes E, Huerta JM, Barricarte A, Amiano P, Sonestedt E, Nilsson LM, Landberg R, Key TJ, Khaw KT, Wareham NJ, Lu Y, Slimani N, Romieu I, Riboli E, Scalbert A. Dietary polyphenol intake in Europe: the European Prospective Investigation into Cancer and Nutrition (EPIC) study. Eur J Nutr. 2016 Jun;55(4):1359-75. doi: 10.1007/s00394-015-0950-x. Epub 2015 Jun 17. PMID 26081647
- [Result] Mohamadpour AH, Ayati Z, Parizadeh MR, Rajbai O, Hosseinzadeh H. Safety Evaluation of Crocin (a constituent of saffron) Tablets in Healthy Volunteers. Iran J Basic Med Sci. 2013 Jan;16(1):39-46. PMID 23638291
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- See also: AIBMR.GRAS Self-determination Inventory Database. Coenzyme Q10. — http://aibmr.com/gras-affirmation-and-the-development-of-functional-foods/
- See also: Centrum — http://labeling.pfizer.com/ShowLabeling.aspx?id=3772
- See also: Omega-3 Fatty Acids — https://medlineplus.gov/druginfo/meds/a607065.html
- See also: Two-Per-Day capsules — http://www.lifeextension.com/Vitamins-Supplements/item02114/Two-Per-Day-Capsules